CLINICAL TRIAL: NCT01449942
Title: Phase I/II Study of EBV-LMP1 Targeted DNAzyme in Nasopharyngeal Carcinoma
Brief Title: Clinical Study of EBV-LMP1 Targeted DNAzyme to Treat Nasopharyngeal Carcinoma
Acronym: NPC-DZ
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Sun lunquan, Director, Center for Molecular Medicine, Central South University, Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSU-863-DZ
Record Dates: First submitted 2011-10-04; First posted 2011-10-10 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; EBV; LMP1
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DZ1 (Experimental): DZ1 group receives DZ1 intratumoral injection in combination with radiation therapy.
  Interventions: Biological: DNAzyme targeting EBV-LMP1 (DZ1); Other: Saline
- Saline (Placebo Comparator): Placebo group receives saline injection in combination with radiation therapy.
  Interventions: Biological: DNAzyme targeting EBV-LMP1 (DZ1); Other: Saline

INTERVENTIONS:
Biological: DNAzyme targeting EBV-LMP1 (DZ1) — DZ1 in saline is administrated by intratumoral injection two hours prior to radiation therapy from week 1 to week 7 on Monday and Thursday. Dosage for each injection is 12 mg in 0.1 mL (200 micrograms per kilogram body weight.
  The radical radiotherapy is given to patients 5 times per week with 2 Gy of each treatment. The entire procedure lasts seven weeks.
Other: Saline — 0.1 mL of saline is administrated by intratumoral injection two hours prior to radiation therapy from week 1 to week 7 on Monday and Thursday.
  The radical radiotherapy is given to patients 5 times per week with 2 Gy of each treatment. The entire procedure lasts seven weeks.

SUMMARY:
The purpose of this study is to determine whether an EBV-LMP1 targeted DNAzyme is effective in radiosensitization of nasopharyngeal carcinoma in combination with standard radiation therapy.

DETAILED DESCRIPTION:
INTRODUCTION Nasopharyngeal carcinoma (NPC) is a serious health problems worldwide, particularly in the southern Chinese population, with an incidence rate ranging from 15 to 50 per 100 000. NPC is an epithelial malignancy with a striking racial and geographic distribution differences. High incidence rates are observed in the southeast Chinese population, and similar rates have been reported in these people wherever they have migrated, including Singapore, Taiwan, and Hong Kong. This incidence is almost 100 fold higher than in white populations. The most unique feature of NPC is its almost universal association with the infection of Epstein-Barr virus (EBV), which is the first human virus identified to be involved in the pathogenesis of several malignancies and has a particularly close association with NPC, as EBV genome can be detected in virtually all NPC cells. While radiotherapy has been the first-line treatments for NPC, radio-resistance remains a significant clinical issue for the NPC radiotherapy. Thus, there is unmet medical needs to discover and develop novel radiosensitizers for NPC therapy.

EBV infection in NPC is classified as type II latent infection in which only EBV nuclear antigen-1(EBNA-1), latent membrane protein-1(LMP1), LMP2, and EBV early RNA (EBER) expressions can be detected. Among these proteins, LMP1 is thought to play a key role in the pathogenesis of NPC. As a 60kD integral membrane protein, LMP1 functions as a constitutively active tumor necrosis factor receptor (TNFR), and contributes to multiple aspects of NPC through activating a number of signaling pathways including nuclear factor NF-κB, activator protein-1(AP-1), and Janus kinase/signal transducer and activator of transcription(JAK/STAT). Activation of NF-kB or AP-1 by LMP1 has been linked to the upregulation of some cellular proteins and inhibition of apoptosis. Depending on the cell types, expression of LMP1 has been shown to play different roles in response to biological and physiological stimulus. It acts as a primary oncoprotein for human cell immortalization and is also shown as the only EBV-coded product that can transform rodent fibroblast cell line, human epithelial cells and keratinocytes.

Given the critical role of viral oncoproteins in transformation and apoptosis, suppression of some viral oncoproteins would provide a sensible strategy to genetically treat NPC. Indeed, antisense oligonucleotides against LMP1 or EBNA1 have been shown to inhibit viral oncoprotein expression, induce apoptosis, and sensitize the EBV-positive cells to cytotoxic agents. Recently, some experimental studies indicated that the RNA interference against LMP1 exhibited an anti-proliferative and anti-metastasis effect in LMP1 expressing NPCs. These results suggested that EBV-encoded LMP1 may present a potential molecular target for treatment of EBV-associated carcinomas.

DNAzymes are synthetic, single-stranded DNA oligonucleotides that can be engineered to bind to their complementary sequence in a target messenger RNA (mRNA) through Watson-Crick base pairing and cleave the mRNA at predetermined phosphodiester linkages. A general model for the DNAzyme has been proposed, and is known as the ''10-23'' model. A ''10-23'' DNAzyme has a catalytic domain of 15 deoxyribonucleotides, flanked by two substrate-recognition domains of seven to nine deoxyribonucleotides at each arm. In vitro analyses showed that this type of DNAzyme could effectively cleave its substrate RNA at purine: pyrimidine junctions under physiological conditions. These agents have been used in a number of in vitro and in vivo applications to inhibit the expression of their target genes and the dependent genes. Their capacity to block development of a diverse range of pathologies in animal models suggests that DNAzymes can be used as therapeutic agents.

To develop EBV-LMP1 targeted DNAzymes for NPC treatment, we showed that the phosphorothioate-modified ''10-23'' DNAzymes specifically targeted at the LMP1 mRNA could significantly down-regulate the expression of LMP1 in a nasopharyngeal carcinoma cell (NPC) and affected the down-stream pathways activated by LMP1, including the NF-κB pathway. It was also demonstrated that suppression of the LMP1 expression by the LMP1-targeted DNAzyme DZ1 could enhance radiosensitivity both in vivo and vitro. Radio-resistance has been one of the impediments in clinical settings for effective cancer therapy, which is thought to be associated with multiple signaling pathways in different cancer types. ATM (ataxia telangiectasia mutated) is a nuclear 350-kDa protein kinase with a carboxylterminal phosphatidylinositol 3-kinase-like kinase domain[1]. It functions as a member of a coordinated system that detects DNA breaks; arrests the cells temporarily at G1, S, or G2 checkpoints; and activates DNA repair. Cells lacking functional ATM protein show increased sensitivity to ionizing radiation (IR) and other genotoxic events. NF-κB (nuclear factor kappa B) can activate a great number of genes involved in stress responses, inflammation, and programmed cell death (apoptosis). P50 homodimers or p50/p65 or p50/c-Rel heterodimers bind to the NF-κB DNA binding sites in the promoter regions of many stress-responsive genes, suggesting a complex gene and physiological regulation network controlled by NF-κB in stress response. The elevated basal NF-κB activity in certain cancers has been linked to tumor resistance to chemotherapy and radiation. Inhibition of NF-κB blocked the adaptive radioresistance. Our studies for the molecular mechanism of the LMP1-DNAzyme mediated radiosensitization revealed that LMP1 activated the ATM expression through the NF-κB pathway and inhibition of LMP1 expression by the DNAzyme attenuated the binding of NF-κB transcription factor to the ATM promoter. Further evidence showed that the radiosensitivity was recovered when the ATM expression was knocked down by siRNA in NPCs. Together, all our data support our hypothesis and provide solid experimental basis for the use of LMP1-targeted DNAzymes as potential radiosensitizers for treatment of the EBV-associated carcinomas.

Toxicological studies in mice showed that no morbidity or mortality was observed in any of the dosing groups during the course of the study (50mg, 100mg, and 200mg/kg). All hematological values and biochemistry results from tests of hepatic and renal function were normal. No microscopic lesion that could be attributed to the modified DNAzyme oligonucleotide treatment was found in liver, spleen and kidney in any groups. After i.v. administration of 100 mg/kg DNAzyme oligonucleotide in mice, the peak plasma concentration of 24.13±2.6μg/ml was achieved. The decrease in plasma concentration of DNAzyme followed a bi-exponential pattern with initial distribution half-life (t1/2α) of 0.18±0.03 h and a terminal half-life (t1/2β) of 2.55±1.0 h, and area under the plasma concentration-time curve (AUC) was 54.17±9.1μg.h/ml.

STUDY DESIGN This study will be a randomized, double-blinded and placebo controlled Phase I/II clinical trial. Forty (40) patients will be randomized to one of two groups of equal size: placebo group receiving saline by intra-tumor injection and standard radiotherapy; or DZ1 group receiving LMP1 DNAzyme (DZ1) and standard radiotherapy. The placebo group will provide the basis for assessment of safety and efficacy of DZ1.

Patients receive placebo or DZ1 injection two (2) hours prior to radical radiation therapy on Monday and Thursday over seven weeks. The radical radiotherapy is given to patients 5 times per week with 2 Gy of each treatment. The entire procedure lasts seven weeks.

All patients will complete the study at 104 weeks post-first injection. The patients will undergo assessment and testing every week in the first seven weeks, then every three months from the weeks 8 to week 104.

The study will include evaluations of safety and tolerability:

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of nasopharyngeal squamous carcinoma
* EBV-LMP1 positive
* Signed Informed Consent Form

Exclusion Criteria:

* Abnormal laboratory results within 45 days prior to study entry
* Participation in any study involving an experimental drug or an experimental medical device in 30 days prior to study entry
* Current pregnancy
* Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Tumor regression rate measured by MRI | Two years
  Tumor growth is measured using MRI weekly from week 1 to week 7, followed by six-monthly measures until week 104.

SECONDARY OUTCOMES:
Tumor vasculature permeability and EBV DNA copies | Two years
  Tumor vasculature permeability is measured using DCE-MRI from week 1 to week 52. EBV DNA copies are measured monthly up to 24 months.EBV cpoies are measured by quantitative PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Lun-Quan Sun, PhD, Principal Investigator — Xiangya Hospital, Central South University, Changsha, China
Locations (1):
- XiangYa Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Yang L, Lu Z, Ma X, Cao Y, Sun LQ. A therapeutic approach to nasopharyngeal carcinomas by DNAzymes targeting EBV LMP-1 gene. Molecules. 2010 Sep 1;15(9):6127-39. doi: 10.3390/molecules15096127. PMID 20877211
- [Background] Lu ZX, Ma XQ, Yang LF, Wang ZL, Zeng L, Li ZJ, Li XN, Tang M, Yi W, Gong JP, Sun LQ, Cao Y. DNAzymes targeted to EBV-encoded latent membrane protein-1 induce apoptosis and enhance radiosensitivity in nasopharyngeal carcinoma. Cancer Lett. 2008 Jul 8;265(2):226-38. doi: 10.1016/j.canlet.2008.02.019. Epub 2008 Mar 18. PMID 18353539
- [Background] Lu ZX, Ye M, Yan GR, Li Q, Tang M, Lee LM, Sun LQ, Cao Y. Effect of EBV LMP1 targeted DNAzymes on cell proliferation and apoptosis. Cancer Gene Ther. 2005 Jul;12(7):647-54. doi: 10.1038/sj.cgt.7700833. PMID 15803142
- [Background] Dass CR, Saravolac EG, Li Y, Sun LQ. Cellular uptake, distribution, and stability of 10-23 deoxyribozymes. Antisense Nucleic Acid Drug Dev. 2002 Oct;12(5):289-99. doi: 10.1089/108729002761381276. PMID 12477279
- [Background] Sun LQ, Cairns MJ, Saravolac EG, Baker A, Gerlach WL. Catalytic nucleic acids: from lab to applications. Pharmacol Rev. 2000 Sep;52(3):325-47. PMID 10977866
- [Background] Cairns MJ, Hopkins TM, Witherington C, Wang L, Sun LQ. Target site selection for an RNA-cleaving catalytic DNA. Nat Biotechnol. 1999 May;17(5):480-6. doi: 10.1038/8658. PMID 10331809
- [Background] Cao Y, DePinho RA, Ernst M, Vousden K. Cancer research: past, present and future. Nat Rev Cancer. 2011 Sep 15;11(10):749-54. doi: 10.1038/nrc3138. PMID 21918542
- [Background] Zheng H, Li LL, Hu DS, Deng XY, Cao Y. Role of Epstein-Barr virus encoded latent membrane protein 1 in the carcinogenesis of nasopharyngeal carcinoma. Cell Mol Immunol. 2007 Jun;4(3):185-96. PMID 17601372
- [Derived] Liao WH, Yang LF, Liu XY, Zhou GF, Jiang WZ, Hou BL, Sun LQ, Cao Y, Wang XY. DCE-MRI assessment of the effect of Epstein-Barr virus-encoded latent membrane protein-1 targeted DNAzyme on tumor vasculature in patients with nasopharyngeal carcinomas. BMC Cancer. 2014 Nov 18;14:835. doi: 10.1186/1471-2407-14-835. PMID 25407966